CLINICAL TRIAL: NCT01772043
Title: Duchenne Muscular Dystrophy Tissue Bank for Exon Skipping
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Sponsor
Other Study IDs: CHAR0312
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: muscular dystrophy; tissue bank
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples with DNA Skin samples Muscle samples (optional)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Duchenne muscular dystrophy

SUMMARY:
We will utilize the Cooperative International Neuromuscular Research Group (CINRG) network to collect and store tissue and blood from patients with Duchenne muscular dystrophy (DMD) with specific genetic mutations within the dystrophin gene that could be treated by antisense oligonucleotide (AO) drugs.

DETAILED DESCRIPTION:
The purpose of this tissue bank is to collect blood and skin samples from participants who are diagnosed with Duchenne muscular dystrophy (DMD) and carry one of nine specific changes in the dystrophin gene. The specific dystrophin changes that we are interested in studying are those that would work with exon-skipping therapies in patients with DMD, specifically deletions of the follow exons: 10-52, 13-50, 29-50, 43-52, 44, 43-50, 45-50, 45-52, 46, 46-47, 46-48, 46-49, 46-51, 46-53, 46-55, 46-60, 47-50, 47-52, 48-50, 49-50, 50, 52, 52-63, 48-52, 49-52, 50-52.

These blood and skin samples will be held in a tissue bank at Carolinas Medical Center for future DMD research.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 and above
* Diagnosis of DMD with a confirmed out-of-frame dystrophin gene deletions that could be corrected by skipping exon 45, 51, or 53 based on past genetic testing.

Exclusion Criteria:

* Investigator assessment of inability to comply with blood and skin sample collection

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Duchenne muscular dystrophy (DMD) is an X-linked recessive disorder caused by mutations in the dystrophin gene. DMD participants over 4 years of age with known mutations that could be targeted by exon skipping therapies will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Tissue Collection | 1 day
  Collection of blood, skin and optional muscle samples

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - University of California Davis, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - Children's National Health System, Washington D.C., District of Columbia
  - Johns Hopkins University School of Medicine, Kennedy Krieger, Baltimore, Maryland
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
- Alberta Children's Hospital, Calgary, Alberta, Canada